CLINICAL TRIAL: NCT02485626
Title: HARBOR Study: Identifying Subgroups With High Cardiovascular Risk in Breast Cancer Survivors
Brief Title: Identifying Subgroups With High Cardiovascular Risk in Breast Cancer Survivors
Acronym: HARBOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: NL49405.031.14
Record Dates: First submitted 2015-06-23; First posted 2015-06-30 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Breast Neoplasms; Cardiovascular Diseases
Keywords: Anthracyclines
MeSH Terms: conditions — Breast Neoplasms; Cardiovascular Diseases | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Consent is obtained from participants to draw blood for DNA-analyses to evaluate whether specific genes modify the risk of treatment-induced cardiovascular disease.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anthracycline treated BC patients: AVL or UMCG patients between the age of 40 - 50 at the time of BC diagnosis and treatment, treated with anthracyclines respectively 5-7 years ago and 10-12 years ago.
  Interventions: Procedure: 2D tissue doppler echocardiography
- Anthracycline naive BC patients: AVL or UMCG patients between the age of 40 - 50 at the time of BC diagnosis and treatment, treated without anthracyclines respectively 5-7 years ago and 10-12 years ago.
  Interventions: Procedure: 2D tissue doppler echocardiography

INTERVENTIONS:
Procedure: 2D tissue doppler echocardiography
  Other Names: laboratory biomarker analyses; vascular ultrasound; strain and strain rate parameters; genetic analysis; questionnaire administration; quality of life assessment; anxiety and depression assessment

SUMMARY:
The purpose of this study is to evaluate the prevalence of (sub)clinical cardiovascular disease, cardiovascular risk factors and metabolic abnormalities among long-term breast cancer survivors treated with or without anthracyclines in order to identify patients at increased risk of developing cardiovascular disease.

DETAILED DESCRIPTION:
Rationale: Breast cancer (BC) incidence is increasing, while mortality from BC is decreasing. Since the life expectancy of BC patients is improving, the evaluation of treatment-associated cardiovascular disease (CVD) in BC survivors is becoming increasingly important. An excess risk of CVD, mainly due to coronary heart disease (CHD), has been observed after radiotherapy (RT) as administered in the 1960s-1980s. Anthracycline-containing CT and trastuzumab are known to induce cardiotoxicity, especially congestive heart failure (CHF). However, the long-term risks of CVD after anthracycline-containing CT, trastuzumab, hormonal therapy (HT) and contemporary RT techniques have hardly been examined. Furthermore, the potential interaction of these treatment modalities has not been well addressed, and there is limited knowledge about the contribution of classic cardiovascular risk factors and the metabolic syndrome to risk and severity of treatment-associated CVD in BC survivors.

Objectives: • to evaluate the prevalence of (sub)clinical CVD, cardiovascular risk factors and metabolic abnormalities among BC survivors treated with and without anthracyclines in two groups at (a) 5 - 7 years and (b) 10 - 12 years after diagnosis;

• to prospectively evaluate changes in prevalence of (sub)clinical CVD, cardiovascular risk factors and metabolic abnormalities after two years in the same patients.

Secondary objectives are to evaluate the predictive role of newly developed markers for CVD and to evaluate the effects of other BC treatment modalities, psychosocial outcomes, endocrine function and menopausal status on the risk of developing (sub)clinical CVD.

Study design: multicenter (AVL and UMCG) cross-sectional cohort study with prospective monitoring of the same cohort.

Study population: female BC survivors treated with and without anthracyclines 5 - 7 and 10 - 12 years ago at the AVL or UMCG, aged 40-50 years at time of therapy.

Main study parameter: the difference in (sub)clinical cardiovascular damage between patients treated with and without anthracyclines, as measured by left ventricular function parameters.

ELIGIBILITY:
Inclusion Criteria:

* early invasive BC (TNM stage I - III);
* diagnosed and/or treated in the AVL or UMCG;
* treated 5 - 7 years or 10 - 12 years ago;
* aged 40-50 years at time of therapy;
* signed written informed consent.

Exclusion Criteria:

* history of RT or CT unrelated to BC;
* current treatment for BC recurrence or second malignancy (including contralateral BC) with the exception of non-melanoma skin cancer or curatively treated carcinoma in situ of the cervix;
* history of cardiac disease (CHF, acute coronary syndrome, coronary revascularization procedure, symptomatic valvular dysfunction, cardiomyopathy or congenital heart defect) before diagnosis and treatment for BC;
* mental disability or psychological condition potentially hampering compliance with the study protocol;
* insufficient understanding of the Dutch language.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited from a large retrospective cohort of BC patients.
Sampling Method: Probability Sample
Enrollment: 628 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | up to 12 years after breast cancer diagnosis
  The main study parameter will be the difference in left ventricular ejection fraction between patients treated with and without anthracyclines.

SECONDARY OUTCOMES:
Diastolic cardiac function | up to 12 years after breast cancer diagnosis
  To compare diastolic cardiac function as measured by tissue doppler echocardiography (E/e' and E/A ratio) in patients treated with and without anthracyclines.
Cardiac deformation | up to 12 years after breast cancer diagnosis
  To compare cardiac deformation as measured by speckle tracking imaging (global longitudial strain, radial strain and circumferential strain) in patients treated with and without anthracyclines.
Biomarker assessment | up to 12 years after breast cancer diagnosis
  To compare levels of several (candidate) cardiovascular biomarkers (NT-proBNP, hs-TnT, CRP) in patients treated with and without anthracyclines.
Intima media thickness and arterial stiffness | up to 12 years after breast cancer diagnosis
  To compare intima media thcikness and arterial stiffness as measured by vascular ultrasound in patients treated with and without anthracyclines.

OTHER OUTCOMES:
Prospective evaluation of changes in LVEF, diastolic cardiac function, cardiac deformation, biomarkers levels, intima media thickness and arterial stiffness after two years in the same patients. | up to 14 years after breast cancer diagnosis
  To compare each outcome of the first and second assessment separately in 1) every patient and 2) between patients treated with and without anthracyclines.

CONTACTS AND LOCATIONS:
Overall Officials: Flora E. van Leeuwen, Prof. dr., Principal Investigator — The Netherlands Cancer Institute
Locations (2):
- Netherlands (2):
  - NKI-AVL, Amsterdam
  - UMCG, Groningen

REFERENCES:
- [Derived] van Ommen-Nijhof A, Jacobse JN, Steggink LC, Lefrandt JD, Gietema JA, van Leeuwen FE, Schaapveld M, Sonke GS. Adjuvant aromatase inhibitor therapy and early markers for cardiovascular disease in breast cancer survivors. Breast Cancer Res Treat. 2022 Dec;196(3):591-602. doi: 10.1007/s10549-022-06714-0. Epub 2022 Oct 1. PMID 36181605